CLINICAL TRIAL: NCT01528917
Title: An Observational Study of the Clinical Characteristics and Disease Progression of Patients With Lysosomal Acid Lipase Deficiency/Cholesteryl Ester Storage Disease Phenotype
Brief Title: An Observational Study of Patients With Lysosomal Acid Lipase Deficiency/Cholesteryl Ester Storage Disease Phenotype
Status: Completed | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LAL-2-NH01
Record Dates: First submitted 2012-02-01; First posted 2012-02-08 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2013-04

CONDITIONS: Cholesterol Ester Storage Disease(CESD); Lysosomal Acid Lipase Deficiency
Keywords: Lysosomal Storage Disease; Late Onset Lysosomal Acid Lipase (LAL) Deficiency; Acid cholesteryl ester hydrolase deficiency, type 2; Acid lipase disease; Cholesterol ester hydrolase deficiency; LAL Deficiency; LIPA Deficiency; Wolman disease
MeSH Terms: conditions — Cholesterol Ester Storage Disease; Wolman Disease; Lysosomal Storage Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a Natural History study to characterize key aspects of the clinical course of late onset Lysosomal Acid Lipase (LAL) Deficiency/ Cholesteryl Ester Storage Disease (CESD).

DETAILED DESCRIPTION:
The objective of this study is to characterize key aspects of the clinical presentation, disease phenotype and progression of patients with late onset Lysosomal Acid Lipase (LAL) Deficiency/ Cholesteryl Ester Storage Disease (CESD) including, but not limited to, age of presentation, onset of hepatomegaly, progression over time of liver function, and stability of lipid abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Patients with late onset LAL Deficiency/ Cholesteryl Ester Storage Disease (CESD) who are 5 years of age or older and have required data points in their medical record

Exclusion Criteria:

* Required data points for inclusion are not available

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with late onset LAL Deficiency/ Cholesteryl Ester Storage Disease (CESD).
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2011-06; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Clinical History Summary | Expected average of 15 years
  Characterize patient demographic data and clinical course of disease using descriptive statistics.

CONTACTS AND LOCATIONS:
Locations (16):
- United States (6):
  - Stanford University, Stanford, California
  - Children's Memorial Hospital, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - Morgan Stanley Children's Hospital of New York-Presbyterian, New York, New York
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Seattle Children's, Seattle, Washington
- Hospital for Sick Kids, Toronto, Canada
- 1st Faculty of Medicine Charles University, Prague, Czechia
- Hôpital Necker-Enfants Malades, Paris, France
- Italy (2):
  - Gaslini Institute, Genoa
  - Regina Margherita Hospital, Turin
- Children's Memorial Health Institute, Warsaw, Poland
- Hopitaux Universitares De Geneve, Geneva, Switzerland
- United Kingdom (3):
  - Birmingham Children's Hospital, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - Salford Royal, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burton BK, Silliman N, Marulkar S. Progression of liver disease in children and adults with lysosomal acid lipase deficiency. Curr Med Res Opin. 2017 Jul;33(7):1211-1214. doi: 10.1080/03007995.2017.1309371. Epub 2017 Apr 3. PMID 28320214
- [Derived] Burton BK, Deegan PB, Enns GM, Guardamagna O, Horslen S, Hovingh GK, Lobritto SJ, Malinova V, McLin VA, Raiman J, Di Rocco M, Santra S, Sharma R, Sykut-Cegielska J, Whitley CB, Eckert S, Valayannopoulos V, Quinn AG. Clinical Features of Lysosomal Acid Lipase Deficiency. J Pediatr Gastroenterol Nutr. 2015 Dec;61(6):619-25. doi: 10.1097/MPG.0000000000000935. PMID 26252914
- See also: Alexion Pharmaceuticals — http://alexion.com/